CLINICAL TRIAL: NCT02734368
Title: A Prospective, Cohort Study of Hyperpolarized 3He MRI in Chronic Obstructive Pulmonary Disease
Status: Terminated | Type: Observational
Why Stopped: The longitudinal goal could not be completed due to CT scans not being performed at baseline.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: COPD-807859
Record Dates: First submitted 2015-05-29; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy non-smokers: Hyperpolarized Helium-3. Amounts adjusted based on subject's total lung capacity
  Interventions: Drug: Hyperpolarized Helium-3
- Asymptomatic smokers: Hyperpolarized Helium-3. Amounts adjusted based on subject's total lung capacity
  Interventions: Drug: Hyperpolarized Helium-3
- COPD subjects: Hyperpolarized Helium-3. Amounts adjusted based on subject's total lung capacity
  Interventions: Drug: Hyperpolarized Helium-3

INTERVENTIONS:
Drug: Hyperpolarized Helium-3

SUMMARY:
The purpose of this study is to determine the MRI characteristics of Chronic Obstructive Pulmonary Disease subjects both at baseline and yearly for a period of 5 years, and to correlate these biomarkers with pulmonary function tests, CT scan, 6 Minute-walk tests, and respiratory questionnaires.

The central hypothesis is that quantitative assessment of the lung through magnetic resonance imaging of hyperpolarized 3He can detect early alterations in structure and function which are precursors to clinically apparent COPD and that these precursors can be used to predict progression of disease earlier and better than established clinical methods.

Novel assessments using 3He MRI will lead to new information about COPD and will be critical for characterizing disease response to therapy. A secondary hypothesis is that a variety of technical improvements in the techniques of hyperpolarized gas MRI will accelerate the translation of this relatively new modality to clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was obtained and documented (after the investigator has given oral and written information about the study to the subject).
* The subject was conscious, co-operative, and agreed to return for the scheduled visits and tests and any visits required to obtain additional safety information.
* The subject's medical history, physical examination (including vital signs, pulse oximetry, PFT's, and 12-lead electrocardiogram [ECG]), and clinical laboratory tests (hematology, serum chemistry) obtained at the screening visit were within acceptable limits for entry into the study, as judged by the investigator.

Exclusion Criteria:

* Subject is <40 or >70 years old
* Subject known to be pregnant
* Subject with a baseline oxygen requirement > 2 l/min via nasal cannula
* Any known contraindication to MRI examination
* Inability to provide informed consent
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed consent
* Active drug or alcohol dependence
* Homelessness or other unstable living situation
* Active drug or alcohol dependence
* Significant co-morbidities such as heart disease, kidney disease, liver disease, hematologic or neurological disease that require continuing treatment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Smoking-Induced Alterations in the Regional Alveolar Oxygen Tension Heterogeneity [Torr] in Smokers Compared to Healthy Controls and COPD Subjects | 2 years from baseline (+- 2 months)
  To measure the specificity and sensitivity of Regional Alveolar Oxygen Tension Heterogeneity in differentiation of healthy smokers from healthy nonsmokers and COPDs
Smoking-Induced Alterations in the Apparent Diffusion Coefficient [cm^2/s] in Smokers Compared to Healthy Controls and COPD Subjects | 2 years from baseline (+- 2 months)
  To measure the specificity and sensitivity of Apparent Diffusion Coefficient in differentiation of healthy smokers from healthy nonsmokers and COPDs
Smoking-Induced Alterations in the Specific Ventilation [unitless] in Smokers Compared to Healthy Controls and COPD Subjects | 2 years from baseline (+- 2 months)
  To measure the specificity and sensitivity of Specific Ventilation in differentiation of healthy smokers from healthy nonsmokers and COPDs

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya R Divgi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.med.upenn.edu/fmig/